CLINICAL TRIAL: NCT05370833
Title: Observation et Analyse Des Effets de la Stimulation transcrânienne à Courant Continu en Milieu Clinique Pour Soulager la Douleur Chronique Chez Les Travailleurs Vieillissants
Brief Title: Transcranial Direct Current Stimulation in Clinical Setting to Reduce Pain in Older Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: CISSS Abitibi-Témiscamingue (Unknown)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-31-2022-4640
Record Dates: First submitted 2022-04-11; First posted 2022-05-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain; Aging
Keywords: transcranial direct current stimulation; physical therapy; work retention
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard protocol (Experimental): 5 tDCS sessions in 1 week
  Interventions: Device: transcranial direct current stimulation
- Enhanced protocol (Experimental): 11 tDCS sessions devised in 4 weeks
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Anodal, 2mA, tDCS session applied on M1 for 20 minutes.

SUMMARY:
Chronic pain is one of the main factors influencing workers' retention at work. Considering that the prevalence of suffering from chronic pain increases with age, older workers are most likely to be absent from work because of their pain.

Transcranial direct current stimulation (tDCS) is a treatment option to reduce chronic pain.

This study aims to document the effect of tDCS on pain and work retention in older workers and to compare the traditional tDCS protocol (5 sessions) with an enhanced protocol (11 sessions).

DETAILED DESCRIPTION:
Chronic pain affects many spheres of the lives of affected individuals and those around them. In Canada, the prevalence of chronic pain is estimated at 15% of adults aged 18 and over. Among seniors, the prevalence of this health problem can reach up to 50% and affect one in two seniors. Chronic pain is one of the leading causes of work disability. In this context, pain reduction remains one of the most effective methods to enable the worker to stay at work. Considering the aging Quebec population, labor needs and the average retirement age which is increasingly postponed, it becomes crucial to take an interest in aging workers and their continued employment.

Transcranial direct current stimulation (tDCS) is a non-invasive neurostimulation method that has shown promise in reducing chronic pain. Recently, several research teams have shown that tDCS has beneficial effects on pain, physical function and social participation in seniors. Despite all these recent advances, very few studies have focused on optimizing tDCS treatment modalities and no studies have focused on the impact of tDCS on return to work or retention. The vast majority of studies using tDCS to reduce pain give one tDCS session per day for 5 consecutive days. This study aims to document the effect of tDCS on pain and work retention in older workers and to compare the traditional tDCS protocol (5 sessions) with an enhanced protocol (11 sessions).

ELIGIBILITY:
Inclusion Criteria:

* To be more than 55 years old
* To have chronic pain
* To have employment relationship
* To have pain that interferes with work tasks

Exclusion Criteria:

- tDCS contraindications (epilepsy, metallic implant in the head, pacemaker, cochlear implant)

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Before tDCS
  0-10 Numerical rating scale
Pain intensity | 1 week
  0-10 Numerical rating scale
Pain intensity | 4 weeks
  0-10 Numerical rating scale
Pain intensity | 4 weeks after the last tDCS session
  0-10 Numerical rating scale
Disability | Before tDCS
  Pain Disability Index
Disability | 1 week
  Pain Disability Index
Disability | 4 weeks
  Pain Disability Index
Disability | 4 weeks after the last tDCS session
  Pain Disability Index
Work role functioning | Before tDCS
  Work Role Functioning Questionnaire
Work role functioning | 1 week
  Work Role Functioning Questionnaire
Work role functioning | 4 weeks
  Work Role Functioning Questionnaire
Work role functioning | 4 weeks after the last tDCS session
  Work Role Functioning Questionnaire
Physical Functioning | Before tDCS
  Brief Pain Inventory
Physical Functioning | 1 week
  Brief Pain Inventory
Physical Functioning | 4 weeks
  Brief Pain Inventory
Physical Functioning | 4 weeks after the last tDCS session
  Brief Pain Inventory
Anxiety | Before tDCS
  Beck anxiety inventory
Anxiety | 1 week
  Beck anxiety inventory
Anxiety | 4 weeks
  Beck anxiety inventory
Anxiety | 4 weeks after the last tDCS session
  Beck anxiety inventory
Depression | Before tDCS
  Beck depression inventory
Depression | 1 week
  Beck depression inventory
Depression | 4 weeks
  Beck depression inventory
Depression | 4 weeks after the last tDCS session
  Beck depression inventory
Impression of change | 1 week
  Patient Global impression of change
Impression of change | 4 weeks
  Patient Global impression of change
Impression of change | 4 weeks after the last tDCS session
  Patient Global impression of change
Central sensitization | Before tDCS
  central sensitization inventory
Central sensitization | 1 week
  central sensitization inventory
Central sensitization | 4 weeks
  central sensitization inventory
Central sensitization | 4 weeks after the last tDCS session
  central sensitization inventory

SECONDARY OUTCOMES:
Recruitment | through study completion, about 2 years
  Feasibility of the study
Security | through study completion, about 2 years
  Feasibility of the study
Intervention | through study completion, about 2 years
  Feasibility of the study

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Leonard, PhD, Principal Investigator — Université de Sherbrooke
Locations (2):
- Canada (2):
  - Clinique régionale de la gestion de la douleur - CISSSAT, Rouyn-Noranda, Quebec
  - Centre de Recherche sur le Vieillissement, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Upon request to the corresponding author
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request